CLINICAL TRIAL: NCT06664710
Title: Evaluation of the Automated Integration of a Robotics and ECochG System for Use With Cochlear Implant Surgery
Acronym: AIMBOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: iotaMotion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: IAR2401
Record Dates: First submitted 2024-10-15; First posted 2024-10-29 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-01

CONDITIONS: Hearing Loss, Sensorineural; Cochlear Implantation
Keywords: cochlear implantation; sensorineural hearing loss; robotics
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (Active Comparator): Use of the iotaSOFT Insertion System and AIM based on Standard of Care
  Interventions: Device: iotaSOFT Insertion System with AIM Control
- Experimental (Experimental): Use of iotaSOFT Insertion System with AIM experimental device
  Interventions: Device: iotaSOFT Insertion System with AIM

INTERVENTIONS:
Device: iotaSOFT Insertion System with AIM — Experimental subjects will receive the iotaSOFT Insertion System with AIM using robotic controlled stop
  Arms: Experimental
Device: iotaSOFT Insertion System with AIM Control — iotaSOFT Insertion System with AIM using standard of care insertion techniques
  Arms: Control

SUMMARY:
Evaluation of the Automated Integration of a Robotics and ECochG System for Use with Cochlear Implant Surgery

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the feasibility and proof of concept of the integration of the AIM System and iotaSOFT Insertion System during cochlear implantation. Study results will help inform the need for future clinical investigations and data collection in the area of ECochG and robotic-assisted cochlear implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Cochlear implant candidate in one or two ears per current FDA indications
2. Sufficient residual hearing to support use of electrocochleography, as determined by the investigator
3. Cochlear implantation using the Advanced Bionics SlimJ electrode array
4. 18 years of age or older at the time of enrollment
5. Willingness to participate in and comply with all requirements of the protocol

Exclusion Criteria:

Contraindications for a CI. 2. Prior cochlear implantation in the ear to be implanted. 3. Cochlear ossification or malformation (including but not limited to dysplasia or common cavity), craniofacial abnormality or any other structural cochlear abnormality that might prevent complete insertion of the electrode array or present an increased risk of aberrant insertion.

4. History of temporal bone fracture that involves the cochlea/internal auditory canal.

5. Retrocochlear etiology (e.g. diagnosis of auditory neuropathy, cochlear nerve deficiency, or lesions of the acoustic nerve or central auditory pathway).

6. Active middle-ear infection or tympanic membrane perforation in the presence of active middle ear disease.

7. Planned or current participation in a clinical study of an investigational device or drug that may impact data collection or outcomes related to this investigation.

8. Additional medical concerns that would prevent participation in evaluations as determined by the investigator.

9. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the procedure and investigational device.

10. Vulnerable subject, as per FDA regulations 21 CFR Parts 50 and 56

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Device Feasibility | Procedure Day 0
  Feasibility of device functionality intraoperatively at the time of cochlear implant surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined based on the results of the study.